CLINICAL TRIAL: NCT04121780
Title: Interventional Study of Growth Hormone Replacement Therapy in Retired Professional Football Players With Growth Hormone Deficiency
Brief Title: Growth Hormone Replacement Therapy for Retried Professional Football Players
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Center for Neurological Studies (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UTN: U1111-1201-5972
Record Dates: First submitted 2019-09-25; First posted 2019-10-10 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: TBI (Traumatic Brain Injury); Concussion, Brain; Sport Injury; Anterior Pituitary Hyposecretion Syndrome; Hypopituitarism; Growth Hormone Deficiency
Keywords: TBI; GHD; Growth Hormone; Norditropin Flexpro; cognition disorders
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion; Hypopituitarism; Dwarfism, Pituitary; Cognition Disorders | interventions — Growth Hormone; Human Growth Hormone; Injections

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled trial with an open-label extension
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: 3-D printing used to design matching cases (covers) for both the drug and placebo autoinjector pens
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Growth Hormone (Experimental): Norditropin® (somatropin [rDNA origin] injection) via FlexPro® 30 mg / 3ml strength auto-injector pens (Novo Nordisk Inc).
  Interventions: Biological: Growth Hormone
- Saline (Placebo Comparator): Saline-placebo via auto-injector pens (Haselmeier Inc).
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Growth Hormone — Daily self-injections by subjects:
  1-year double-blind phase; 6-month open-label extension for those who received placebo during the double-blind phase
  Other Names: Norditropin® (somatropin [rDNA origin] injection)
  Arms: Growth Hormone
Other: Placebo — Daily self-injections by subjects:
  1-year double-blind phase
  Arms: Saline

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel-group trial with an open-label extension to evaluate the efficacy of growth hormone (GH) on cognitive functions of retired professional football players with growth hormone deficiency (GHD).

DETAILED DESCRIPTION:
GHD is the most common anterior pituitary abnormality after traumatic brain injury (TBI). It can occur as a result of either direct pituitary or indirect hypothalamic injury. Sports-related repetitive head trauma might induce pituitary dysfunction, and in particular, isolated GHD. Growth hormone replacement therapy (GHRT) has long been known to have a beneficial effect on body composition and exercise capacity. However, it has recently been shown that GHRT also benefits the brain. The primary objective of the current study is to assess the effect of GH on memory, executive function and attention domains of cognitive function in GHD- professional football players with TBI. The study will also utilize the adult growth hormone deficiency assessment (AGHDA) questionnaire, quantitative electroencephalogram (QEEG) and magnetic resonance imaging (MRI) techniques, respectively, to measure the quality of life (QoL), electrical activity and structural changes in the brain that may correspond to cognitive deficits.

ELIGIBILITY:
Inclusion Criteria:

* The subject is willing to provide a signed and dated informed consent indicating that he understands the purpose and procedures required for the study and is willing to participate in the study.
* Former NFL player
* At least one year since retirement from football
* Less than 76 years of age
* Diagnosis of GHD on clinical grounds by a neurologist and an endocrinologist GHD

Exclusion Criteria:

* History of pre-existing brain disease other than concussion or TBI
* History of a premorbid disabling condition that interferes with outcome assessments
* Contraindication to GH therapy
* Type I and II Diabetes mellitus
* Active malignant disease
* Acute critical illness, heart failure, or acute respiratory failure
* Subjects who are deficient in cortisol, testosterone or thyroid at screening will be excluded until hormone abnormalities have been corrected.

Ages: 18 Years to 76 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2019-10-08 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Cognitive functions- Working Memory | From baseline to 1-year post-treatment
  To assess change in working memory from base line to 1 yr post-treatment. Working memory will be reported as an index score based on scaled scores for the digit span subtest and symbol span subtest. Index scores have a mean of 100 and a standard deviation of 15. The typical range of index score is 45 to 155. Higher scores reflect better functioning. The scaled scores have a mean of 10 and a standard deviation of 3. Scores range from 1 to 19. Higher scores reflect better functioning.
Cognitive functions- Processing Speed | From baseline to 1-year post-treatment
  To assess change in Processing Speed from baseline to 1 yr post-treatment. Processing speed will be reported as an index score based on scaled scores of digit symbol subtest and symbol search subtest. Index scores have a mean of 100 and a standard deviation of 15. The typical range of index score is 45 to 155. Higher scores reflect better functioning. The scaled scores have a mean of 10 and a standard deviation of 3. Scores range from 1 to 19. Higher scores reflect better functioning.
  Trail Making Test A will also be used to assess processing speed. Reported as T-score. Higher scores reflect better performance.
Cognitive functions- Executive Function. | From baseline to 1-year post-treatment
  To assess change in Executive Function from baseline to 1 yr post-treatment. Trail Making Test B and verbal fluency (letter and category) will be used to assess executive function. Reported as T-score. T scores have a mean of 50 and a standard deviation of 10. Scores range from 13 to 87. Higher scores reflect better performance.
Cognitive functions- Verbal learning and memory | From baseline to 1-year post-treatment
  To assess change in Verbal learning and memory from baseline to 1 yr post-treatment. California verbal learning test will be used to assess this outcome measure. Reported as a standard score with a mean of 0 and a standard deviation of 1. Scores range from -0.5 to +5.0. Higher scores reflect better performance.
Cognitive functions- ANAM ( Automated Psychological Assessment Metrics) | From baseline to 1-year post-treatment
  To assess change in ANAM from baseline to 1 yr post-treatment. ANAM Test System- Core Battery will be used to assess this outcome measure. Reported as a standard score

SECONDARY OUTCOMES:
Quality of Life Assessment of Growth Hormone Deficiency in Adults | One year (from baseline to 1-year post-treatment)
  This measure includes a scale: It is based on the Adult Growth Hormone Deficiency Assessment (AGHDA) QoL questionnaire. It consists of 25 yes/no questions. Score ranges from 0-25 with number of "yes" responses indicating score. A score of 8 or higher is typical of untreated adult GH deficiency. Treatment, on an average, results in a decrease of 2.5 to 3 points on the scale at one year
Change in QEEG Markers- power spectra | One year (from baseline to 1-year post-treatment)
  Spectral markers include delta (1-5-2.5 Hz), theta (3.5-7.5 Hz), alpha (7.5-12.5 Hz), alpha 1 (7.5-10.0 Hz), alpha 2 (10.0-12.5 Hz), beta 1 (12.5- 25.0 Hz) , beta 2 (25.0-35.0 Hz), gamma (35.0- 50.0 Hz). The power will be averaged over all electrode sites as absolute and relative power.
Change in QEEG Markers- Connectivity Measures | One year (from baseline to 1-year post-treatment)
  Connectivity measures will include Pearson product moment correlation for the time series and coherence, phase synchronization and phase lag.
MRI | One year (from baseline to 1-year post-treatment)
  To assess changes in volumetric MRI measurements and diffusion tensor imaging (DTI) measurements
Change in Physical function- Peak O2 consumption (Vo2 max) | One year (from baseline to 1-year post-treatment)
  Measured in units of liters per minute.
Change in Physical function- Maximum grip strength | One year (from baseline to 1-year post-treatment)
  Measured in pounds using the CAMRY Digital Hand Dynamometer
Change in Physical function- Isokinetic knee extension peak torque | One year (from baseline to 1-year post-treatment)
  Measured using the Cybex II isokinetic dynamometer. The maximum torque is recorded in ft-lbs of force
Change in Physical function-DEXA measure | One year (from baseline to 1-year post-treatment)
  Percent body fat and lean mass by limb and trunk
Adverse events | One year (from baseline to 1-year post-treatment)
  To assess the incidence and severity of adverse events

OTHER OUTCOMES:
MR imaging analysis of hypothalamus and pituitary | One year (from baseline to 1-year post-treatment)
  for diagnosis of GHD or multiple anterior pituitary hormone deficiencies in GHD - professional football players with TBI

CONTACTS AND LOCATIONS:
Overall Officials: Randall R Benson, MD, Principal Investigator — Vice President and Medical Director
Locations (1):
- Center for Neurolgoical Studies (CNS), Dearborn, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benson RR, Gattu R, Sewick B, Kou Z, Zakariah N, Cavanaugh JM, Haacke EM. Detection of hemorrhagic and axonal pathology in mild traumatic brain injury using advanced MRI: implications for neurorehabilitation. NeuroRehabilitation. 2012;31(3):261-79. doi: 10.3233/NRE-2012-0795. PMID 23093454
- [Background] Benson RR, Meda SA, Vasudevan S, Kou Z, Govindarajan KA, Hanks RA, Millis SR, Makki M, Latif Z, Coplin W, Meythaler J, Haacke EM. Global white matter analysis of diffusion tensor images is predictive of injury severity in traumatic brain injury. J Neurotrauma. 2007 Mar;24(3):446-59. doi: 10.1089/neu.2006.0153. PMID 17402851
- [Background] Falleti MG, Maruff P, Burman P, Harris A. The effects of growth hormone (GH) deficiency and GH replacement on cognitive performance in adults: a meta-analysis of the current literature. Psychoneuroendocrinology. 2006 Jul;31(6):681-91. doi: 10.1016/j.psyneuen.2006.01.005. Epub 2006 Apr 18. PMID 16621325
- [Background] Deijen JB, de Boer H, Blok GJ, van der Veen EA. Cognitive impairments and mood disturbances in growth hormone deficient men. Psychoneuroendocrinology. 1996 Apr;21(3):313-22. doi: 10.1016/0306-4530(95)00050-x. PMID 8817729
- [Background] Deijen JB, de Boer H, van der Veen EA. Cognitive changes during growth hormone replacement in adult men. Psychoneuroendocrinology. 1998 Jan;23(1):45-55. doi: 10.1016/s0306-4530(97)00092-9. PMID 9618751
- [Background] Kelestimur F, Tanriverdi F, Atmaca H, Unluhizarci K, Selcuklu A, Casanueva FF. Boxing as a sport activity associated with isolated GH deficiency. J Endocrinol Invest. 2004 Dec;27(11):RC28-32. doi: 10.1007/BF03345299. PMID 15754728
- [Background] Kelly DF, Chaloner C, Evans D, Mathews A, Cohan P, Wang C, Swerdloff R, Sim MS, Lee J, Wright MJ, Kernan C, Barkhoudarian G, Yuen KC, Guskiewicz K. Prevalence of pituitary hormone dysfunction, metabolic syndrome, and impaired quality of life in retired professional football players: a prospective study. J Neurotrauma. 2014 Jul 1;31(13):1161-71. doi: 10.1089/neu.2013.3212. Epub 2014 May 8. PMID 24552537
- [Background] High WM Jr, Briones-Galang M, Clark JA, Gilkison C, Mossberg KA, Zgaljardic DJ, Masel BE, Urban RJ. Effect of growth hormone replacement therapy on cognition after traumatic brain injury. J Neurotrauma. 2010 Sep;27(9):1565-75. doi: 10.1089/neu.2009.1253. PMID 20578825
- [Background] Reimunde P, Quintana A, Castanon B, Casteleiro N, Vilarnovo Z, Otero A, Devesa A, Otero-Cepeda XL, Devesa J. Effects of growth hormone (GH) replacement and cognitive rehabilitation in patients with cognitive disorders after traumatic brain injury. Brain Inj. 2011;25(1):65-73. doi: 10.3109/02699052.2010.536196. Epub 2010 Nov 30. PMID 21117918
- [Background] Moreau OK, Cortet-Rudelli C, Yollin E, Merlen E, Daveluy W, Rousseaux M. Growth hormone replacement therapy in patients with traumatic brain injury. J Neurotrauma. 2013 Jun 1;30(11):998-1006. doi: 10.1089/neu.2012.2705. Epub 2013 Jun 5. PMID 23323993
- [Background] Devesa J, Reimunde P, Devesa P, Barbera M, Arce V. Growth hormone (GH) and brain trauma. Horm Behav. 2013 Feb;63(2):331-44. doi: 10.1016/j.yhbeh.2012.02.022. Epub 2012 Mar 1. PMID 22405763